CLINICAL TRIAL: NCT01465867
Title: Selenium Supplementation Treatment in Euthyroid Pregnant Women With Autoimmune Thyroid Disease: Effects on Obstetrical Complications
Brief Title: Selenium Supplementation in Pregnancy
Acronym: Serena
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea M. Isidori, Principal Investigator, Clinical Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Sel-01
Record Dates: First submitted 2011-11-02; First posted 2011-11-07 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Pregnancy; Infertility; Auto-immune Thyroiditis
Keywords: Selenium; Pregnancy; Auto-immune thyroiditis; Post-partum thyroiditis; Miscarriage; Pre-eclampsia; Implantation and Pregnancy rate; Infertility
MeSH Terms: conditions — Infertility; Postpartum Thyroiditis; Abortion, Spontaneous; Pre-Eclampsia | interventions — Selenium; Sugars; Methods; phospholamban; Thyroxine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Selenium (Experimental)
  Interventions: Dietary Supplement: Selenium
- Sugar Pill Placebo (Placebo Comparator)
  Interventions: Other: Sugar Pill Placebo
- Selenium + L-Thyroxine (LT4) (Experimental)
  Interventions: Other: Selenium + L-Thyroxine (LT4)
- Sugar Pill Placebo + L-Thyroxine (LT4) (Experimental)
  Interventions: Other: Sugar Pill Placebo + L-Thyroxine (LT4)

INTERVENTIONS:
Dietary Supplement: Selenium — 83 micrograms of selenium (in the form of selenium methionine) in tablet form taken orally daily for all the length of pregnancy and for 3-6th month after labour
  Other Names: Intervention I (Se)
  Arms: Selenium
Other: Sugar Pill Placebo — Placebo supplements in the same capsule as selenium. 1 tablet daily for all the length of pregnancy and for 3-6th month after labour.
  Other Names: Intervention II (Plb)
  Arms: Sugar Pill Placebo
Other: Selenium + L-Thyroxine (LT4) — 83 micrograms of selenium (in the form of selenium methionine) in tablet form taken orally daily for all the length of pregnancy and for 3-6th month after labour
  + LT4 taken orally daily according to the dose required(in women already receiving it or needing of start it)
  Other Names: Intervention III (Se+LT4)
  Arms: Selenium + L-Thyroxine (LT4)
Other: Sugar Pill Placebo + L-Thyroxine (LT4) — Placebo supplements in the same capsule as selenium. 1 tablet daily for all the length of pregnancy and for 3-6th month after labour
  + LT4 taken orally daily according to the dose required(in women already receiving it or needing of start it)
  Other Names: Intervention IV (Plb + LT4)
  Arms: Sugar Pill Placebo + L-Thyroxine (LT4)

SUMMARY:
Serum levels of isolated anti-thyroperoxidase (TPOab) and anti-thyreoglobulin (Tgab) autoantibodies are strongly associated with an increased risk of miscarriage and premature deliveries in euthyroid pregnant women. Replacement of thyroxine (LT4) or other supplementations in euthyroid-Ab positivity during pregnancy has not been established. The development of a safe and effective intervention that modulates inappropriate inflammatory responses could be a very important component of prevention against adverse health outcomes during pregnancy.

The anti-oxidant Selenium (Se) suppresses autoimmune destruction of thyrocytes and at daily dose of 200 mcg and 100 mcg decreases titers of serum TPOAb and TgAb also in Se-non-deficient patients with autoimmune thyroiditis (AIT).

The use of Se in AIT has been shown to reduce the incidence of postpartum thyroiditis and hypothyroidism.

Women with recurrent pregnancy loss had lower Se levels and Se deficiency has been implicated in the pathogenesis of AIT and in the impairment of T/B cell-mediated immunity.

The purpose of the present study is performed to establish the effect of Se supplementation in euthyroid women with AIT (pregnant and in whom embryo transfer is expected within 60 days) on Ab trend, thyroid function and structure, implantation rates, pregnancy rates, pregnancy outcome and number of obstetrical, fetal and neonatal complications.

DETAILED DESCRIPTION:
Adverse outcomes, postpartum thyroid dysfunction and permanent hypothyroidism have been associated with isolated TPOab positivity in euthyroid pregnant women.

In areas with severe selenium deficiency there is a higher incidence of thyroiditis due to a decreased activity of selenium-dependent glutathione peroxidase activity within thyroid cells. Selenium-dependent enzymes also have several modifying effects on the immune system. Therefore, even mild selenium deficiency may contribute to the development and maintenance of autoimmune thyroid diseases.

Selenium substitution exerts anti-inflammatory and anti-oxidant activities. Se could represents an important supplementation in euthyroid women with AIT in order to improve thyroid function and structure and to prevent obstetrical adverse events related to autoimmune diseases and reactive oxygen species, such as recurrent miscarriage and pre-eclampsia.

The aim of this study is to document the effects of Selenium Supplementation with and without L-thyroxine (LT4) in euthyroid women with AIT, during pregnancy.

This protocol will evaluate the trend of TPOab and Tgab, selenium concentration, thyroid volume and echogenicity, nodule formation and number of adverse effects that affect the mother (during and after pregnancy), the fetus, the infant and the heath service, needing to elucidate the nature of the emerging associations.

The study also aims to assess the impact of Selenium Supplementation on implantation rate and pregnancy rate in women with transfer planned within the next 60 days.

This is designed as a phase IV study on treatment with a cohort size of pregnant women and women in whom embryo transfer is expected within 60 days with TSH value into the normal range (0.4-2.5 mUI/mL) and Tgab and/or TPOab positivity. We have performed two randomizations arms: Randomization arm A will include women LT4 replacement-free that will take Selenium or Placebo and Randomization arm B will include women already under LT4 replacement that will take Selenium or Placebo. Patients included in Randomization A will move into Randomization B, if TSH increases above 2.5 mUI/mL during pregnancy.

Pregnant women with TSH > 2.5 mU/mL at time 0 will begin (or will adjust) LT4 replacement and will be included in Randomization arm B.

Accounting for a 30% drop off, a total enrolment of 150 patients is planned. Patients will be randomized at time 0 (10°± 2 weeks of gestation). Follow-up visits will take place at weeks 14 ± 2, 24 ± 2, 32 ± 2, 36 ± 2 weeks, and between months 3° and 6° after labour. An optional visit could be done 12 months after labor. Plasma and serum monitoring of thyroid hormones, Tgab, TPOab, Se concentration, Selenoproteins and cytokines, thyroid US, SF12 questionnaire will be made at all the follow-up visits. At visit 3 (24 ± 2 weeks) patients will optionally do the OGTT). Gestational, obstetrical, maternal, fetal, and infant anamnestic data will be taken, during the follow up visits and at labour.

The long-term objective is to identify a safe and easily administered supplementation that improves:

1. implantation and pregnancy rates in infertile women Tgab and/or TPOab positives
2. maternal and fetal complication in pregnant euthyroid women Tgab and/or TPOab positives.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with 10°± 2 weeks of gestation
* women in whom embryo transfer is expected within 60 days
* euthyroid women (0.4 μIU/ml < TSH < 2.5 μIU/ml), positive for TPOab and/or TgAb, not assuming LT4 replacement
* euthyroid women (0.4 μIU/ml < TSH < 2.5 μIU/ml), positive for TPOab and/or TgAb under LT4 replacement (to maintain TSH within the control range).
* women with TSH > 2.5 μIU/ml positive for TPOab and/or TgAb, not assuming LT4 replacement (requiring the beginning of LT4 replacement)
* women with TSH > 2.5 μIU/ml positive for TPOab and/or TgAb, under LT4 replacement (requiring an adjustment of LT4 replacement)

Exclusion Criteria:

* use of dietary supplements containing selenium in the previous 4 months;
* use of antidepressive/psychotic drugs, amiodarone, propanolol, lithium, cytokines;
* history of hyperthyroidism positive anti-thyrotropin ab;
* previous partial or total thyroidectomy;
* known fetal anomaly;
* known infections (PID, HIV, HCV) and mola hydatidoses;
* chronic renal failure;
* uncontrolled hypertension;
* uterine malformation;
* history of medical and metabolic complication such as heart disease or diabetes;
* previous embryo transfer failed within last 3 months;
* miscarriage within last 3 months;
* gestational diabetes in previous pregnancies.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2012-04; Primary Completion 2017-06 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Changes in TPOab and/or Tgab | 0 and 14 ± 2, 24 ± 2, 32± 2, 36± 2 weeks; and between 3° and 6° month after labour; and optionally 12° after labour
  TPOab and Tgab titers will be measured using a ECLIA kit. Plasma selenium concentration will also be measured

SECONDARY OUTCOMES:
Changes in thyroid volume and echogenicity | 0 and 14 ± 2, 24 ± 2, 32± 2, 36± 2 weeks; and between 3° and 6° month after labour; and optionally 12° after labour
  Also changes in thyroid nodules diameters and/or nodules formation will be measured by Ultrasonographic (US) imaging
Changes in thyroid hormones (TSH, FT4, FT3) | 0 and 14 ± 2, 24 ± 2, 32± 2, 36± 2 weeks; and between 3° and 6° month after labour; and optionally 12° after labour
Evaluation of Maternal risks | From the date of randomization until the date of first documented event
  Pre-eclampsia (gestational hypertension: systolic pressure ≥140 mmHg or diastolic blood pressure ≥ 90 mmHg [Korotkoff V] on ≥ 2 occasions after 20 weeks gestation), Miscarriage, Placental Abruption, Abruption, Gestational hypertension, Breech presentation at birth, Preterm birth (< 37 weeks gestation), Symptomatic hypothyroidism, Preterm labour, Postpartum haemorrhage, Postpartum depression, Postpartum Thyroiditis, Maternal death
Evaluation of Infant risks | From the date of labour until the date of the first documented event
  Small for gestational age, Admission to special care, Cretinism, Jaundice requiring phototherapy, Poor feeding, Constipation, Hoarse cry, Lethargy, Hypotonia, Macroglossia, Umbilical hernia
Changes in of quality of life | 0 and 14 ± 2, 24 ± 2, 32± 2, 36± 2 weeks; and between 3° and 6° month after labour; and optionally 12° after labour
  Quality of life will be measured by questionnaire SF12
Evaluation of Health Services: | from the date of admission until the date of discharge
  Maternal length of hospital stay (days), Neonatal length of hospital stay (in days), Cost of services
Changes in the selenium-dependent antioxidant enzyme glutathione peroxidase | 0, 24 ± 2, 36± 2 weeks; and 6 months after labour
  Glucose, Vitamin B-12, folate, methionine, albumin and cytokines will be also measured in serum
Changes in implantation and pregnancy rates | From the date of embryo transfer until the date of documented progression
  Clinical implantation rate (IR) and pregnancy rate (PR)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Isidori, MD, PhD, Principal Investigator — Department of Experimental Medicine, Section of Clinical Pathophysiology and Endocrinology, "Sapienza" University of Rome
Locations (11):
- Italy (11):
  - Azienda ospedaliero-universitaria Careggi, Florence
  - Istituto Auxologico Italiano, Milan
  - Ospedale Maggiore Policlinico, Milan
  - University Federico II, Naples
  - University "Piemonte Orientale, A. Avogadro", Novara
  - Torvergata University of Rome - Ospedale S. Eugenio, Rome
  - European Hospital, Rome
  - Ospedale S. Giovanni Calibita Fatebenefratelli, Rome
  - Department of Experimental Medicine, "Sapienza" University of Rome, Rome
  - Department of Gynecological/Obstetric/Urological Sciences, "Sapienza" University of Rome, Rome
  - Dpt of Experimental Medicine, Rome